CLINICAL TRIAL: NCT00687076
Title: Effect of Lipid Modification on Peripheral Arterial Disease After Endovascular Intervention ("The ELIMIT Trial")
Brief Title: Effectiveness of Intensive Lipid Modification Medication in Preventing the Progression of Peripheral Arterial Disease (The ELIMIT Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christie Ballantyne, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1400; R01HL075824 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Endovascular Intervention; MRI; Ultrasound; Cholesterol Medications; High Cholesterol; Peripheral Arterial disease; Claudication; Leg Pain; Niaspan; Extended Release Niacin; Zetia; Ezetimibe; Simvastatin; Zocor; Atorvastatin; Lipitor
MeSH Terms: conditions — Peripheral Arterial Disease; Hypercholesterolemia; Intermittent Claudication | interventions — Ezetimibe; Niacin; Simvastatin; Standard of Care; Aspirin; Clopidogrel; Angioplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive standard of medical care and treatment with intensive lipid modification using a statin plus Ezetimibe and Niaspan.
  Interventions: Drug: Ezetimibe; Drug: Niaspan; Drug: Statin therapy; Behavioral: Standard care; Drug: Aspirin; Drug: Clopidogrel; Procedure: Percutaneous transluminal angioplasty (PTA)
- 2 (Active Comparator): Participants will receive standard of medical care and treatment with standard lipid modifying medications plus placebo Ezetimibe and placebo Niaspan.
  Interventions: Drug: Statin therapy; Behavioral: Standard care; Drug: Aspirin; Drug: Clopidogrel; Drug: Placebo Niaspan; Drug: Placebo Ezetimibe; Procedure: Percutaneous transluminal angioplasty (PTA)

INTERVENTIONS:
Drug: Ezetimibe — Daily dose of 10 mg of Ezetimibe
  Other Names: Zetia
  Arms: 1
Drug: Niaspan — Daily dose of 1500 mg of Niaspan
  Other Names: Extended release niacin
  Arms: 1
Drug: Statin therapy — Daily dose of 40 mg of Simvastatin (If unable to tolerate Simvastatin, participants will take a daily dose of Atorvastatin.)
  Other Names: Zocor; Liptior
Behavioral: Standard care — Standard of medical care for PAD
Drug: Aspirin — Daily dose of 325 mg of aspirin
Drug: Clopidogrel — Daily dose of 75 mg of clopidogrel for 3 months or as recommended by the primary care physician
  Other Names: Plavix
Drug: Placebo Niaspan — Daily dose of 1500 mg of placebo Niaspan
  Arms: 2
Drug: Placebo Ezetimibe — Daily dose of 10 mg of placebo Ezetimibe
  Arms: 2
Procedure: Percutaneous transluminal angioplasty (PTA) — Participants who have not had an endovascular intervention in the 3 months before study entry will undergo PTA to mechanically open the artery blockages. This procedure will involve the inflation and deflation of a small balloon to open the blocked artery. Additionally, participants may have a metal mesh tube called a stent placed in the blocked area if deemed necessary by their physicians.
  Other Names: Endovascular intervention

SUMMARY:
Peripheral arterial disease (PAD) occurs when arteries become narrowed or hardened because of a build-up of plaque or fat deposits. PAD develops most often in arteries in the legs, which can result in reduced blood flow to the legs and feet, occasionally causing leg pain and fatigue. Early identification of PAD and treatment with lifestyle changes or medications can help to keep legs healthy and lower risk for heart attack and stroke, but endovascular or surgical procedures may be necessary for people with severe PAD. Even after endovascular intervention, PAD symptoms must be continually monitored to prevent the development and progression of blockages in the arteries. The best approach for monitoring symptoms is still undetermined. This study will compare the effectiveness of an intensive combination of lipid modifying medications versus standard lipid modifying medications in treating people with significant PAD who have had an endovascular intervention.

DETAILED DESCRIPTION:
PAD occurring in the legs is a serious disease that affects about 8 million people in the United States. A person's risk for PAD increases with age but can also be raised by smoking or having diabetes, high blood pressure, high cholesterol, or heart disease. Symptoms of PAD may include leg cramps or pain while walking, foot pain while resting, and skin wounds or ulcers on feet and toes. However, because only about one in three people with PAD knows to seek treatment for these symptoms, many end up with advanced disease that requires significant medical intervention, such as an endovascular or other surgical procedure to open the blocked arteries. While these procedures are helpful in treating people with severe PAD, lifestyle modifications and certain medications are also needed for long-term management of PAD and improved quality of life. An intensive combination of lipid modifying medications may be superior to standard lipid modifying medications in reducing PAD-associated risk factors and improving overall health in people with PAD. This study will compare the effectiveness of an intensive combination of lipid modifying medications versus standard lipid modifying medications in preventing blockages and re-narrowing of arteries in people with significant PAD who have had an endovascular intervention.

Participation in this study will last a minimum of 2 years and a maximum of 5 years. All participants will first undergo baseline assessments that will include a medical history, vascular and physical exam, electrocardiograph (EKG), magnetic resonance imaging (MRI) scan, 3D ultrasound, blood pressure measurement test in the legs, treadmill walking distance test, urine test, blood draw, and questionnaires. A portion of the blood draw will be used for DNA analysis and genetic testing.

Participants who have not had an endovascular intervention in the 3 months before study entry will undergo a standard of care percutaneous transluminal angioplasty (PTA) procedure. First these, participants will complete a series of clinical review assessments that will include a review of social, vascular, and clinical history. Next, they will undergo the PTA procedure, which will involve the inflation and deflation of a small balloon in the area of the blocked artery. Additionally, participants may have a metal mesh tube called a stent placed in the blocked area, if deemed necessary by their physicians.

All participants will then be assigned randomly to receive standard care plus an intensive combination of lipid modifying medications (Simvastatin, Plavix, aspirin, Ezetimibe, and Niaspan) or standard lipid modifying medications with placebo (Simvastatin, Plavix, aspirin, placebo Ezetimibe, and placebo Niaspan). Participants will take their assigned medications daily for 24 months. Follow-up visits will occur at Day 10; Week 6; and Months, 6, 12, and 24 after beginning the study medications. During follow-up visits, participants will repeat the baseline assessments and the clinical review assessments from the pre-PTA visit. The Week 6 follow-up visit will include only a blood draw, questionnaires, and the clinical review assessments. Participants will also be contacted by phone to check their status every 2 to 3 months during treatment and every 6 months after treatment for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with calf claudication and described as life style limiting
* Objective evidence of peripheral artery disease (PAD): Ankle brachial index less than 0.9 OR other hemodynamic or imaging modalities confirming significant PAD
* Baseline imaging reveals superficial femoral artery (SFA) disease starting at least 5 cm from the origin of the SFA
* Agrees to be available for follow-up and is able to participate in all study testing procedures
* Weight and/or body characteristics that will allow testing with MRI
* No known contraindication to lipid lowering agents
* Serum creatinine level less than 2.5 mg/dL
* Scheduled to undergo or has already undergone an endovascular intervention of a de novo lesion in the SFA with an anticipated result that would satisfy hemodynamic stability OR is medically managed and does not require an intervention at this time
* Compressible arteries (if not, has toe brachial index [TBI] less than 0.7)
* Has/had an A, B, C lesion amendable to a catheter based therapy (prior bypass is acceptable)

Exclusion Criteria:

* Non-atherosclerotic disease that is responsible for claudication
* Unstable cardiac disease (e.g., unstable angina, heart attack within the 30 days before study entry, uncontrolled coronary heart failure, poorly controlled hypertension [systolic blood pressure greater than 180 mmHg and/or diastolic blood pressure greater than 100 mmHg], ventricular arrhythmias)
* Pancreatitis
* Documented hypercoagulable state
* Clinically severe diabetic neuropathy
* Rest pain, gangrene, or tissue loss
* Active peptic ulcer disease or a recent gastrointestinal bleed that would prohibit the use of an anti-platelet (aspirin/Plavix)
* Untreated or unsuccessfully controlled psychiatric disease
* Chronic hepatic disease determined by aspartate transaminase (AST) and/or alanine transaminase (ALT) more than 3 times upper limit of normal (ULN) and/or total bilirubin more than 2 times ULN
* Creatine phosphokinase (CPK) more than 3 times ULN (may be repeated once before patient is excluded)
* Active gout symptoms or a uric acid level greater than 1.3 times ULN
* Untreated hypothyroidism
* Allergy to Plavix, nickel, titanium, niacin, Ezetimibe, statins, or their derivatives
* Participated in another interventional study within the 30 days before study entry
* Scheduled to undergo planned synchronous bilateral percutaneous transluminal angioplasty (PTA) procedures
* Requires an above the ankle amputation
* Scheduled to undergo elective surgery within 30 days after the PTA procedure
* Has an implanted pacemaker, defibrillator, neural stimulator, brain clip, insulin pump, cochlear implant, or any other predetermined radiographic finding that would exclude MRI testing
* Has claustrophobia that would prevent MRI testing
* Recent drug or alcohol abuse history (less than 6 months before study entry) or is currently using or abusing excessive alcohol or drugs (excessive alcohol will be defined as greater than 14 drinks per week)
* Past recipient of a cardiac, kidney, liver, lung, or other organ transplant (skin grafts are acceptable)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2004-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie M. Ballantyne, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Lumsden AB, Rice TW, Chen C, Zhou W, Lin PH, Bray P, Morrisett J, Nambi V, Ballantyne C. Peripheral arterial occlusive disease: magnetic resonance imaging and the role of aggressive medical management. World J Surg. 2007 Apr;31(4):695-704. doi: 10.1007/s00268-006-0732-y. PMID 17345122
- [Result] Brunner G, Yang EY, Kumar A, Sun W, Virani SS, Negi SI, Murray T, Lin PH, Hoogeveen RC, Chen C, Dong JF, Kougias P, Taylor A, Lumsden AB, Nambi V, Ballantyne CM, Morrisett JD. The Effect of Lipid Modification on Peripheral Artery Disease after Endovascular Intervention Trial (ELIMIT). Atherosclerosis. 2013 Dec;231(2):371-7. doi: 10.1016/j.atherosclerosis.2013.09.034. Epub 2013 Oct 16. PMID 24267254
- [Result] Saunders J, Nambi V, Kimball KT, Virani SS, Morrisett JD, Lumsden AB, Ballantyne CM, Dong JF; ELIMIT Investigators. Variability and persistence of aspirin response in lower extremity peripheral arterial disease patients. J Vasc Surg. 2011 Mar;53(3):668-75. doi: 10.1016/j.jvs.2010.08.029. Epub 2011 Jan 12. PMID 21227624
- See also: Click here for more information on peripheral arterial disease — http://www.nhlbi.nih.gov/health/dci/Diseases/pad/pad_what.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Triple Therapy: Participants will receive standard of medical care and treatment with intensive lipid modification using a statin plus Ezetimibe and Niaspan.
  Ezetimibe: Daily dose of 10 mg of Ezetimibe
  Niaspan: Daily dose of 1500 mg of Niaspan
  Statin therapy: Daily dose of 40 mg of Simvastatin (If unable to tolerate Simvastatin, participants will take a daily dose of Atorvastatin.)
  Standard care: Standard of medical care for PAD
  Aspirin: Daily dose of 325 mg of aspirin
  Clopidogrel: Daily dose of 75 mg of clopidogrel for 3 months or as recommended by the primary care physician
  Inclusion criteria were life-style-limiting claudication consistent with Fontaine Stage IIa/IIb or angiographically confirmed Trans-Atlantic Inter-Society Consensus A-C lesions in the SFA.
- Mono Therapy: Participants will receive standard of medical care and treatment with standard lipid modifying medications plus placebo Ezetimibe and placebo Niaspan.
  Statin therapy: Daily dose of 40 mg of Simvastatin (If unable to tolerate Simvastatin, participants will take a daily dose of Atorvastatin.)
  Standard care: Standard of medical care for PAD
  Aspirin: Daily dose of 325 mg of aspirin
  Clopidogrel: Daily dose of 75 mg of clopidogrel for 3 months or as recommended by the primary care physician
  Placebo Niaspan: Daily dose of 1500 mg of placebo Niaspan
  Placebo Ezetimibe: Daily dose of 10 mg of placebo Ezetimibe
  Inclusion criteria were life-style-limiting claudication consistent with Fontaine Stage IIa/IIb or angiographically confirmed Trans-Atlantic Inter-Society Consensus A-C lesions in the SFA.
Period: Overall Study
Arm/Group | Triple Therapy | Mono Therapy
Started | 51 | 51
Completed | 19 | 21
Not Completed | 32 | 30

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were compared using analysis of variance, chi-square tests. Multilevel statistical models were used to analyze the primary outcome. Complete baseline characteristics were availabe for 95 patients. Between randomization and baseline visit, 1 patient withdrew from study, and 6 patients declined blood collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Therapy | Mono Therapy | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (7.8) | 63.9 (7.1) | 63.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 43 | 46 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 4 | 17
  White | 32 | 44 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Effect of Intensive Lipid Modification Medication Therapy on Progression of Atherosclerosis and Restenosis of Femoral Arteries Measured Using High Resolution Magnetic Resonance Imaging (MRI) to Examine the Femoral Artery for Progression of Atherosclerosis
Description: The primary outcome variable was the change in superficial femoral artery (SFA) wall volume over 24-months, as determined by MRI. The 24-month changes in SFA lumen and SFA total vessel volumes were also analyzed.
  Analysis details: A total of 102 patients were randomized. 87 patients completed baseline MRI. Between randomization and the baseline visit, 1 patient withdrew from the study, 8 patients opted out from baseline imaging, and 6 additional patients declined blood collection at baseline. The multilevel models (primary endpoint) used all available imaging data (n=91), including patients who only completed baseline imaging (n=20) or completed at least 2 imaging visits other than baseline (n=4).
Time Frame: Measured at baseline and 24 Months
Population: Multilevel models were used to describe changes over time in the MRI outcome variables and to compare the drug therapy groups. The advantage of multilevel models is the capability to use data with missing or irregularly timed observations, due to death or loss to follow-up, on the outcome variable.
Measure: Mean (Standard Error); unit: mm^3, at 24-months
Arm/Group | Triple Therapy | Mono Therapy
Number analyzed (Participants) | 45 | 46
mm^3, at 24-months | 58.1 (5.5) | 60.5 (5.1)

2. Secondary Outcome: Change in Total Cholesterol (mg/dl) From Baseline to Month 12
Description: Lipids: Total cholesterol (mg/dl); Lipid Data at 12-Months (change from baseline) [mg/dl].
Time Frame: Measured at baseline and 12 months
Population: All values are medians and interquartile range (IQR). P-values were calculated with the KruskaleWallis rank test.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Triple Therapy | Mono Therapy
Number analyzed (Participants) | 47 | 48
mg/dl | -30.0 [-63 to -1] | -7.5 [-30.5 to 8.0]

ADVERSE EVENTS:
Time Frame: Major adverse events were reported to and assessed by the Data and Safety Monitoring Board (DSMB).
Arm/Group | Triple Therapy | Mono Therapy
All-Cause Mortality (participants affected / at risk) | 4/47 | 4/48
Serious Adverse Events (participants affected / at risk) | 7/47 | 4/48
Other Adverse Events (participants affected / at risk) | 10/47 | 8/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Therapy (N=47) | Mono Therapy (N=48)
Myocardial infarction (Cardiac disorders) | 3 | 1
Major stroke (Cardiac disorders) | 2 | 2
Coronary revascularization (Cardiac disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Therapy (N=47) | Mono Therapy (N=48)
Blood Glucose Adverse Events (Endocrine disorders) | 10 | 8 — Patients with Blood Glucose Adverse Events (excluding Baseline; hyperglycemic adverse events: Blood Glucose > 180 mg/dl ) or Adverse Events of HbA1c > 10%.

LIMITATIONS AND CAVEATS:
MRI was performed in the distal SFA. Ethnicity which was not part of the randomization protocol differed significantly between mono- and triple-therapy groups. The attrition rate was high in ELIMIT. ELIMIT was not powered to assess clinical outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No